CLINICAL TRIAL: NCT01339494
Title: Arginine Flux and Nitric Oxide Production in Patients With MELAS Syndrome and the Effect of Arginine and Citrulline Supplementation
Brief Title: Nitric Oxide Production in MELAS Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Fernando Scaglia, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-24783
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: MELAS Syndrome
MeSH Terms: conditions — MELAS Syndrome | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arginine supplementation (Active Comparator): Oral L-arginine supplementation will be administered to subjects with MELAS for 48 hours at a dose of 10 grams per M2 per day. Arginine will be given every 4 hours.
  Interventions: Dietary Supplement: Arginine and citrulline supplementations
- citrulline supplementation (Active Comparator): Oral L-citrulline supplementation will be administered to subjects with MELAS for 48 hours at a dose of 10 grams per M2 per day. Citrulline will be given every 4 hours
  Interventions: Dietary Supplement: Arginine and citrulline supplementations

INTERVENTIONS:
Dietary Supplement: Arginine and citrulline supplementations — Arginine or citrulline will be given orally at dose of 10 grams per meter square body surface area per day divided every 4 hours.

SUMMARY:
Introduction

Baylor College of Medicine and Texas Children's Hospital are recruiting individuals with MELAS syndrome for a clinical study. MELAS syndrome is a mitochondrial disease; patients with this disease have muscle weakness and often develop brain strokes, where blood does not flow normally to different parts of the brain. It is believed that these strokes could be due to decreased production of nitric oxide, a naturally occurring compound important for normal blood vessel function. Nitric oxide is made from arginine and citrulline that are normally found in our bodies.

What is the purpose of this study? The purpose of this study is to measure nitric oxide in individuals with MELAS and see if giving arginine or citrulline will increase the formation of nitric oxide. Nitric oxide is thought to be helpful in preventing strokes. Therefore, if arginine and/or citrulline are shown to increase the formation of nitric oxide, they could be used to prevent or treat the strokes in patients with MELAS syndrome.

DETAILED DESCRIPTION:
What does the study involve? Individuals with MELAS syndrome will be admitted twice to the General Clinical Research Center (GCRC) at Texas Children's Hospital. Each time they will stay for five days, during which a special diet will be provided. Nitric oxide production will be measured by stable isotopes infusion technique that involves placing small tubes in veins (IV catheter), blood sampling, and injecting a harmless stable isotope. Stable isotopes are forms of normal compounds that can be measured accurately. They are not radioactive and there are no known risks to giving them; they are already part of your body in small amounts.

During the first admission nitric oxide levels will be measured, then arginine supplementation will be provided for 48 hours, after which nitric oxide levels will be re-measured to determine the effect of arginine supplementation. During the second admission, the effect of citrulline supplementation will be measured.

Who can participate in the study? Adults or children affected with MELAS syndrome and carrying the DNA change that causes the condition (3243 A>G mutation) can participate. Adults without MELAS disease will be recruited to participate as control subjects.

How to get more information? Subjects interested in participation or getting more information can contact Dr. Ayman El-Hattab at email: elhattab@bcm.edu, office phone: 832-822-4289, cell phone: 646-660-5666, or pager: 832-824-7243 (5523).

ELIGIBILITY:
Inclusion Criteria:

1. Age from 3 - 65 years
2. Clinical diagnosis of MELAS syndrome
3. Carrying the m.3243A>G mutation

Exclusion Criteria:

1. Having acute or chronic disease or physical disability that will interfere with the ability to undergo the study procedures
2. Being pregnant

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in nitric oxide production | Nitric oxide production will be measured at baseline before supplementation and after 48 hours of arginine or citrulline supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Scaglia, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes the data have been made available to